CLINICAL TRIAL: NCT06761898
Title: A Phase 1, Open-label, Randomized, Crossover Study to Investigate the Relative Bioavailability of Two Tablet Formulations and the Effect of Food on the Pharmacokinetics of a Single Oral Dose of BGB-43395 in Healthy Participants
Brief Title: A Study of Different Forms of BGB-43395 and Food Effect in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BGB-43395-103
Record Dates: First submitted 2024-12-31; First posted 2025-01-07 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers
Keywords: BGB-43395; Relative Bioavailability; Effect of Food; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Relative Bioavailability (Experimental): Participants will receive a single dose of each formulation of BGB-43395 in separate periods across various sequences.
  Interventions: Drug: BGB-43395
- Part 2: Food Effect (Experimental): Participants will receive three doses of the selected formulation of BGB-43395 under fasted, low-fat, or high-fat conditions in separate periods across various sequences.
  Interventions: Drug: BGB-43395

INTERVENTIONS:
Drug: BGB-43395 — Administered orally as solid dispersion tablet or salt tablet
  Arms: Part 1: Relative Bioavailability
Drug: BGB-43395 — Administered orally as solid dispersion tablet or salt tablet
  Arms: Part 2: Food Effect

SUMMARY:
Study to determine the relative bioavailability of BGB-43395 solid dispersion tablet compared to salt tablet in healthy adult participants in Part 1 and the effect of food on the selected BGB-43395 formulation solid dispersion tablet or salt tablet in healthy adult participants in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, of any race, between 18 and 65 years of age
* Body mass index between 18.0 and 32.0 kg/m2, inclusive
* In good health, as determined by no clinically significant findings from medical history
* Able to comprehend and are willing to sign the ICF and abide by the study restrictions

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator or designee
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, as determined by the investigator or designee.
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair are allowed)
* Confirmed systolic blood pressure >140 or <90 mmHg, diastolic blood pressure >90 or <50 mmHg, or pulse rate >100 or <40 beats per minute. If any parameter is out of range, measurements should be repeated twice. Participants will be excluded if the average of the 3 measurements are outside of the corresponding reference range.
* History of prolonged QT interval/QT interval corrected for heart rate, with QTcF >450 ms for males and >470 ms for females.
* History or current diagnosis of diabetes, with a HbA1c ≥6.5% or fasting blood glucose level ≥126 mg/dL at screening alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin >1.5 × upper limit of normal (ULN) (except for participants with Gilbert's syndrome, where total bilirubin should not be >2 × ULN) at screening and check-in.
* eGFR <90 mL/min/1.73 m2 (Chronic Kidney Disease Epidemiology Collaboration (CKD EPI) 2021)
* Hemoglobin <lower limit of normal (LLN), white blood cell count <LLN, absolute neutrophil count <LLN, or platelet count <LLN at screening and check-in.
* Positive hepatitis panel and/or positive human immunodeficiency virus test.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2025-01-14 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Part 1 and 2: Area Under the Concentration-time Curve from Time 0 Extrapolated to Infinity (AUC0-∞) | PK is assessed on days 1-15 in Part 1 and Days 1- 22 for part 2
Part 1 and 2: Area Under the Concentration-time Curve from Time 0 to the Time of the Last Quantifiable Concentration (AUC0-tlast) | PK is assessed on days 1-15 in Part 1 and Days 1- 22 for part 2
Part 1 and 2: Maximum Observed Concentration (Cmax) | PK is assessed on days 1-15 in Part 1 and Days 1- 22 for part 2
Part 1 and 2: Time of the Maximum Observed Concentration (Tmax) | PK is assessed on days 1-15 in Part 1 and Days 1- 22 for part 2
Part 1 and 2: Apparent Terminal Elimination Half-life (t1/2) | PK is assessed on days 1-15 in Part 1 and Days 1- 22 for part 2
Part 1 and 2: Apparent Total Clearance (CL/F) | PK is assessed on days 1-15 in Part 1 and Days 1- 22 for part 2
Part 1 and 2: Apparent Volume of Distribution (Vz/F) | PK is assessed on days 1-15 in Part 1 and Days 1- 22 for part 2

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Approx 38 days in Part 1 and 45 days in part 2
Number of participants with clinically significant laboratory values | Approx 38 days in Part 1 and 45 days in part 2
Number of participants with clinically significant electrocardiogram (ECG) results | Approx 38 days in Part 1 and 45 days in part 2
Number of participants with clinically significant vital sign measurements | Approx 38 days in Part 1 and 45 days in part 2

CONTACTS AND LOCATIONS:
Overall Officials: Study Director Study Director, Study Director — BeiGene
Locations (1):
- Fortrea Cru, Daytone Beach, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
URL: https://www.beigenemedical.com/medical-information-request